CLINICAL TRIAL: NCT07159997
Title: Accuracy OF Rail Sign at Detection Of Placenta Accreta at The Second And the Third Trimester Of Pregnancy By Ultrasound Scanning
Brief Title: Accuracy of Rail Sign at Detection of PAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rehab Zakria Ahmed, Rehab zakaria Ahmed, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med--25-8-5MS
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Placenta Previa Complete Centralis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pregnant femsles with placenta previa (Experimental)
  Interventions: Diagnostic Test: Accuracy of rail sign by ultrasound st diagnosis placent previa

INTERVENTIONS:
Diagnostic Test: Accuracy of rail sign by ultrasound st diagnosis placent previa — Accuracy of rail sign by ultrasound at derection of PAS

SUMMARY:
Accuracy OF Rail Sign at Detection Of Placenta Accreta At The second And the Third Trimester Of Pregnancy By Ultrasound Scanning

ELIGIBILITY:
Inclusion Criteria:

* pregnant femsles with placenta previa

Exclusion Criteria:

* primigravida

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant femsles with placenta previa
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of rail sign by ultrasound at detection PAS | Intraoperative
Accuracy of rail sign at diagnosis of PAS by ultrasound | Inyaroperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided